CLINICAL TRIAL: NCT01049802
Title: Evaluation of Therapeutic Effects of Navigation-guided 1 Hz rTMS Administered to the Contralesional Hemisphere in Patients With Stroke
Brief Title: Contrastim Stroke Trial
Acronym: ContraStim
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Nexstim Ltd (Industry)
Responsible Party: Principal Investigator, Richard Harvey, Medical Director of Stroke Rehabilitation, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NR-001
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Stroke
Keywords: stroke; hemiplegia; TMS
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): Experimental subjects will receive subthreshold or suprathreshold rTMS to contralesional hemisphere for up to 20 minutes at 1 Hz followed by task oriented arm and hand therapy to affected limb.
  Interventions: Device: Repetititve transcranial magnetic stimulation
- Sham rTMS (Placebo Comparator): Subject will receive sham rTMS to contralesional hemisphere for up to 20 minutes followed by task-oriented arm and hand rehabilitation to affected limb
  Interventions: Device: Repetititve transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetititve transcranial magnetic stimulation — 1 Hz rTMS to contralesional hemisphere in patients with stroke

SUMMARY:
This is a prospective randomized controlled feasibility study to determine whether navigation guided repetitive transcranial magnetic stimulation (rTMS) to the healthy hemisphere in patients with subacute stroke has a beneficial effect when given concurrently with task-oriented motor rehabilitation of the arm and hand. Navigation guided rTMS requires a structural MRI scan for targeting stimulation and therefore structural MRI will be performed on all subjects. In addition the study intends to determine whether measures of motor tract integrity (MTI) assessed by navigated brain stimulation (NBS) and MRI diffusion tensor imaging can be used to clarify prognosis of motor recovery and to monitor progress with rehabilitation. 30 subjects with ischemic or hemorrhagic stroke 3-9 months prior to enrollment and with residual upper limb hemiplegia will be randomized to receive either 1 Hz rTMS to the contralesional hemisphere for 30 minutes 3 times a week for 6 weeks along with rehabilitation therapy or sham rTMS to the contralesional hemisphere for 30 minutes 3 times a week for 6 weeks along with rehabilitation therapy. Primary outcome is improvement on the Action Research Arm Test, a measure of arm and hand function in people with stroke. Outcomes will be measured immediately post treatment, and at 3 months and 6 months post treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES To determine whether NBS guided 1Hz rTMS targeting the motor representation areas of hand muscles on the healthy brain hemisphere has a beneficial effect on the motor recovery of the corresponding stroke-affected muscles when combined with standardized task-oriented motor rehabilitation.

SECONDARY OBJECTIVES

1. To determine whether motor evoked potentials (MEPs) can be elicited from paretic and/or plegic muscles in patients with stroke using navigated TMS (eXimia NBS) and targeting the anatomical cortical areas representing the affected muscles.
2. To determine the correlation between existing MEPs, other TMS parameters and the clinical deficits of limb function.
3. To determine the prognostic value of MEPs and other TMS parameters in predicting motor recovery after stroke
4. To determine the diagnostic value of MEPs and other TMS parameters in monitoring the response to rehabilitation
5. To assess safety by capturing all Serious Adverse Events during both single pulse and rTMS delivery

STUDY PROCEDURES

The purpose of the study including risks and benefits will be explained to potential participants who will then be asked to sign an informed consent form. Potential participants will be screened for inclusion and exclusion criteria

The study will be performed in 2 parts. In part 1 Nexstim eXimia NBS will be utilized for neuronavigation and a third party TMS will be used for delivering the rTMS. In part 2 Nexstim eXimia NBS will be utilized together with Nexstim eXimia TMS for delivering the rTMS. Part 2 will commence once the patients participating in Part 1 have undergone the study visit 22 (see 5.1 below).

15 patients will be recruited to part 1 and 15 patients for part 2 (6 additional subjects will be recruited assuming a 20% drop out rate)

In part 1 of the study 10 subjects will be randomized to rTMS treatment and 5 subjects will be randomized to sham rTMS. Of the 10 rTMS treatment subjects, 5 will be given stimulation protocol A and 5 will be given stimulation protocol B, described below. In part 2, either stimulation protocol A or B will be chosen for continue study based on predetermined outcome criteria. In part 2, 10 subjects will receive this chosen rTMS treatment and 5 subjects will receive sham rTMS.

The study will consist of 24 study visits with the addition of 4 additional visits as needed to complete outcome assessments.

VISIT SCHEDULE

The study will be performed over 24 to 28 sessions:

1. Visit 1(Screening visit): Baseline = 3-9 months after the stroke. The purpose of this visit is to obtain informed consent for the study (if not previously obtained) and to screen subjects for inclusion and exclusion criteria.
2. Visit 2: Baseline assessment. The purpose of this visit is to establish the baseline of injury, motor status and NBS parameters (Hand motor mapping and motor tract integrity, both hemispheres - see appendix A). Subjects will also undergo a structural MRI. The subject will then be randomized to either rTMS or to sham treatment. The baseline visit may if necessary take place on 2 separate days.
3. Visits 3-21: During these visits the patient will undergo standardized task-oriented motor rehabilitation of the hand. In addition the patient will receive the rTMS therapy according to the protocol of the group she/he was randomized into during visit 1. The visits will take place during a 6 week period, three visits per week. During each week the visits will take place each on a separate day and a maximum of two visits will take place on consecutive days. During the first visit of each week (visits 3, 6, 9, 12, 15 and 18) in addition to the rTMS and task-oriented motor rehabilitation, the patient will undergo measurement of NBS parameters (Motor tract integrity, both hemispheres).
4. Visit 22: End of the task-oriented motor rehabilitation. The purpose of the visit is to establish the extent of recovery that has occurred during the rehabilitation. The visit will take place 3-5 days after the last rTMS/rehabilitation session and includes functional motor testing and evaluation of NBS parameters (Hand motor mapping and motor tract integrity, both hemispheres). 1-2 visits may be needed to complete assessment.

5) Visit 23: 1 month after the end of the rehabilitation therapy. The purpose of the visit is to determine whether any changes in motor function or NBS parameters have occurred within 1 month of ending therapy. The assessment includes functional motor testing and evaluation of NBS parameters (Hand motor mapping and motor tract integrity, both hemispheres). 1-2 visits may be needed to complete assessment.

6) Visit 24: 6 months after end of the rehabilitation therapy. The purpose of this visit is to determine the long-term rehabilitation success. The assessment includes functional motor testing and evaluation of NBS parameters (Hand motor mapping and motor tract integrity, both hemispheres. In patients experience a new stroke or TIA during this time, only the data prior to the event will be used in the analysis. 1-2 visits may be needed to complete assessment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* An ischemic or hemorrhagic stroke suffered 3-9 months prior to the study
* no other known brain abnormalities by history or by structural MRI
* A one-sided stroke resulting in upper extremity paresis
* A Chedoke Arm and Hand Activity Inventory score of 3-6 for the affected limb

Exclusion Criteria:

* Implanted metallic parts of implanted electronic devices, including pacemakers, defibrillators, or implant medication pump
* Pregnant or trying to become pregnant
* History of alcohol abuse, illicit drug use or drug abuse or significant mental illness
* any history of epilepsy
* Any condition that would prevent the subject from giving voluntary informed consent
* An implanted brain stimulator
* Aneurysm clip or other metal in body
* Enrolled or plans to enroll in an interventional trial during this study
* Scalp wounds or infections
* Claustrophobia precluding MRI
* A fixed contraction deformity in the affected limb
* Excessive spasticity as indicated by the Modified Ashworth Spasticity (MAS) Scale >2/4 in the affected limb
* previous stroke with residual deficits (TIAs not a reason for exclusion)
* premorbid (retrospective) modified Rankin Scale (mRS) score ≥2 of any aetiology
* a concurrent progressive neurologic disorder, acute coronary syndrome, severe heart disease (NYHA Classification > 3), or other major medical condition
* confirmed or suspected lower-limb fracture preventing mobilization
* patients requiring palliative care
* patients undergoing any other occupational therapy than what is provided in the study
* A recent injection of botulinum toxin to the affected upper limb in the last 3 months, or the need of an injection of botulinum toxin anytime during the study period and follow up
* Ataxia as measured by a score > 1 on item 7 (limb ataxia) of the NIH stroke scale
* Severe aphasia as measured by a score of > 2 on item 9 (best language) of the NIH stroke scale
* Severe neglect as measured by a score of 2 on item 11 (extinction and inattention) of the NIH stroke scale

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Harvey, MD, Principal Investigator — The Rehabilitation Institute of Chicago; Jarmo Laine, MD, PhD, MBA, Study Director — Nexstim Ltd
Locations (1):
- The Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: The Rehabilitation Institute of Chicago — http://www.ric.org
- See also: Nexstim Ltd. — http://www.nexstim.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Contralesional rTMS With Arm Rehabilitation: Experimental subjects will receive subthreshold or suprathreshold rTMS to contralesional hemisphere for up to 20 minutes at 1 Hz followed by task oriented arm and hand therapy to affected limb.
  repetitive transcranial magnetic stimulation to contralesional hemisphere: 1 Hz rTMS to contralesional hemisphere in patients with stroke
- Sham Contralesional rTMS Plus Arm Rehabilitation: Subject will receive sham rTMS to contralesional hemisphere for up to 20 minutes followed by task-oriented arm and hand rehabilitation to affected limb
  repetitive transcranial magnetic stimulation to contralesional hemisphere: 1 Hz rTMS to contralesional hemisphere in patients with stroke
Period: Overall Study
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 8 | 23
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Full Range); unit: years] | 59.0 [22 to 90] | 48.1 [20 to 74] | 55.3 [20 to 90]
Gender [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 12 | 5 | 17
Fugl-Meyer Score [Mean (Standard Deviation); unit: units on a scale] — Upper extremity Fugl-Meyer Score measures of motor impairment in hemiplegic upper limb of patients with stroke. The scoring follows the natural progression of motor recovery as defined by Twitchell (Brain. 1951; 64:443-480). The score was developed by Axel Fugl-Meyer and it has been validated (Scand J Rehab Med. 1975; 7:13-31; Stroke. 2009; 40: 1386-1391). The scale ranges 0-66 with 66 representing normal motor function and 0 representing no movement. There are 33 movement items each scored 0 (cannot perform), 1 (peforms partially), 2 (performs flawlessly)
  units on a scale | 23.8 (10.2) | 31.5 (15.3) | 26.4 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Fugl-Meyer Score
Description: Upper extremity Fugl-Meyer Score measures of motor impairment in hemiplegic upper limb of patients with stroke. The scoring follows the natural progression of motor recovery as defined by Twitchell (Brain. 1951; 64:443-480). The score was developed by Axel Fugl-Meyer and it has been validated (Scand J Rehab Med. 1975; 7:13-31; Stroke. 2009; 40: 1386-1391). The scale ranges 0-66 with 66 representing normal motor function and 0 representing no movement. There are 33 movement items each scored 0 (cannot perform), 1 (peforms partially), 2 (performs flawlessly)
Time Frame: Baseline, post treatment, 1 month, 6 months
Population: 6 month outcome is the primary endpoint. 1 data point is missing from the treatment arm at 6 month follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 23.8 (10.2) | 31.5 (15.3)
  Post treatment | 31.9 (14.6) | 37 (18.4)
  1 month | 32.8 (14.9) | 36.1 (18.1)
  6 month | 37.6 (17.3) | 38.6 (16.5)
Statistical Analysis 1: Comparison: Contralesional rTMS With Arm Rehabilitation vs Sham Contralesional rTMS Plus Arm Rehabilitation; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Action Research Arm Test
Description: The ARAT is a measure of upper limb dexterity and is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from:
  * 3: Performs test normally
  * 2: Completes test, but takes abnormally long or has great difficulty
  * 1: Performs test partially
  * 0: Can perform no part of test Range is 0-57 with higher scores relating to better upper limb dexterity
Time Frame: Baseline, post treatment, 1 month, 6 months
Population: 1 data point is missing from treatment arm at both 1 week and 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 20.9 (15.7) | 26.9 (21.2)
  Post treatment | 28.8 (18.5) | 32.5 (21.7)
  1 month | 28.6 (18.8) | 31.3 (19.7)
  6 month | 32.4 (20.2) | 35.5 (18.6)
Statistical Analysis 1: Comparison: Contralesional rTMS With Arm Rehabilitation vs Sham Contralesional rTMS Plus Arm Rehabilitation; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

3. Secondary Outcome: Stroke Impact Scale
Description: The SIS is a quality of life questionnaire designed for stroke survivors. It is a 59 item measure
  * 8 domains assessed:
    * Strength (4 items)
    * Hand function (5 items)
    * ADL/IADL (10 items)
    * Mobility (9 items)
    * Communication (7 items)
    * Emotion (9 items)
    * Memory and thinking (7 items)
    * Participation/Role function (8 items)
  * Each item is rated in a 5-point Likert scale in terms of the difficulty the patient has experienced in completing each item
  * Summative scores are generated for each domain, scores range from 0-100
Time Frame: Baseline, post treatment, 1 month, 6 months
Population: 1 data point is missing from treatment arm a 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 62.4 (10.5) | 63.6 (14.8)
  Post treatment | 74.2 (17.3) | 75.1 (14.7)
  1 month | 70.8 (12.0) | 74.1 (15.6)
  6 month | 74.5 (12.5) | 78.2 (12.2)
Statistical Analysis 1: Comparison: Contralesional rTMS With Arm Rehabilitation vs Sham Contralesional rTMS Plus Arm Rehabilitation; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

4. Secondary Outcome: Chedoke Arm Assessment
Description: A 7 point scale of motor recovery scored separately for arm. 7 is good motor recovery and 1 is no movement.
Time Frame: Screening, baseline, weekly, post treatment, 1 month, 6 months
Population: 1 data point is missing in treatment arm at 6 month post
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 3.35 (0.58) | 4.1 (1.19)
  Post treatment | 4.05 (1.15) | 5.0 (1.7)
  1 month | 4.4 (1.39) | 4.8 (1.69)
  6 month | 4.79 (1.62) | 5.3 (1.77)
Statistical Analysis 1: Comparison: Contralesional rTMS With Arm Rehabilitation vs Sham Contralesional rTMS Plus Arm Rehabilitation; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

5. Secondary Outcome: NIH Stroke Scale
Description: A composite scale derived from the Toronto Stroke Scale, the Oxbury Initial Severity Scale, the Cincinnati Stroke Scale and the Edinburgh-2 Coma Scale
  * 15 items assessing severity of impairment in LOC, ability to respond to questions and obey simple commands, papillary response, deviation of gaze, extent of hemianopsia, facial palsy, resistance to gravity in the weaker limb, plantar reflexes, limb ataxia, sensory loss, visual neglect, dysarthria and aphasia severity
  * Items are graded on a 3 or 4 point ordinal scale; 0 equates no impairment
  * Scores range from 0 - 42. Higher scores indicate greater severity.
  * Stroke severity may be stratified on the basis of NIHSS scores as follows (Brott et al, 1989):
    * Very Severe: >25
    * Severe: 15 - 24
    * Mild to Moderately Severe: 5 - 14
    * Mild: 1 - 5
Time Frame: Screening, baseline, post treatment, 1 month, 6 months
Population: 1 data point missing from treatment arm at 6 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 4.1 (1.55) | 3.3 (1.95)
  Post treatment | 3.15 (1.46) | 2.5 (1.58)
  1 month | 3.6 (1.7) | 2.3 (1.42)
  6 month | 2.58 (1.61) | 2.7 (1.34)
Statistical Analysis 1: Comparison: Contralesional rTMS With Arm Rehabilitation vs Sham Contralesional rTMS Plus Arm Rehabilitation; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Contralesional rTMS With Arm Rehabilitation | Sham Contralesional rTMS Plus Arm Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/10
Other Adverse Events (participants affected / at risk) | 6/20 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contralesional rTMS With Arm Rehabilitation (N=20) | Sham Contralesional rTMS Plus Arm Rehabilitation (N=10)
Hospitalization (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contralesional rTMS With Arm Rehabilitation (N=20) | Sham Contralesional rTMS Plus Arm Rehabilitation (N=10)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Fall (General disorders) | 2 (2) | 2 (2)
Blood pressure instability (Cardiac disorders) | 3 (4) | 0 (0)
Floaters in visual field (Eye disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Active group included combination of two types of active rTMS. Data was intended purely for pilot purposes to estimate sample size for a larger multicenter trial (the NICHE clinical trial).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No